CLINICAL TRIAL: NCT02688179
Title: Neuroinflammation and Postoperative Delirium in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Sponsor
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: 160032
Record Dates: First submitted 2016-02-05; First posted 2016-02-23 (Estimated); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Delirium; Cardiac Surgery
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cardiac surgery patients

SUMMARY:
Up to 50% of patients over 60 years old develop postoperative delirium following cardiac surgery. Delirium increases morbidity and mortality, and may lead to long-term cognitive impairment similar to patients with a diagnosis of Alzheimer's disease. The underlying mechanisms behind delirium are not understood, and therefore the current prevention and treatment strategies are inadequate. Several hypotheses exist for the pathophysiology of delirium, one of which is the role of neuroinflammation. The stress associated with high-risk procedures such as cardiac surgery may lead to systemic inflammation causing endothelial dysfunction and disruption of the blood brain barrier (BBB). When this occurs, the brain is susceptible to neuronal injury via neuroinflammation after which a state of delirium may ensue. To characterize the mechanisms of neuroinflammation in delirium, the investigators will explore the biomarkers most closely linked to each step of the proposed pathway.

DETAILED DESCRIPTION:
Aim 1a. Test the hypothesis that endothelial injury is associated with delirium. The investigators hypothesize that endothelial dysfunction is associated with an increased incidence of delirium after cardiac surgery. To test this hypothesis, the investigators will measure biomarkers from subjects undergoing cardiac surgery. Blood samples from three time points [baseline, upon arrival to the intensive care unit (ICU), and postoperative day 1 (POD1)] will be analyzed and compared between patients that did and did not develop postoperative delirium.

Aim 1b. Test the hypothesis that BBB disruption is associated with delirium. The investigators hypothesize that disruption in the BBB is associated with an increased incidence of delirium after cardiac surgery. To test this hypothesis, the investigators will measure levels of biomarkers at baseline, upon arrival to the ICU, and on POD1.

Aim 1c. Test the hypothesis that neuronal injury is associated with delirium. The investigators hypothesize that neuronal injury is associated with an increased incidence of delirium after cardiac surgery. To test this hypothesis, the investigators will measure levels of biomarkers at baseline, upon arrival to the ICU, and on POD1.

ELIGIBILITY:
Inclusion Criteria:

* open heart surgery

Exclusion Criteria:

* acute coronary syndrome with troponin leak or unrelenting angina
* liver dysfunction (transaminases 2x normal)
* history of myopathy or liver dysfunction on prior statin therapy
* use of potent CYP3A4 inhibitors such as antifungal azoles, macrolide antibiotics, HIV protease inhibitors, and nefazodone.
* pregnancy or breast feeding
* cyclosporine use
* dialysis
* history of kidney transplant
* fibrate users who cannot stop fibrate use

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 undergoing open heart surgery
Sampling Method: Non-Probability Sample
Enrollment: 630 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
change in endothelial dysfunction | baseline, postoperative day 0, postoperative day 1
  biomarker of endothelial dysfunction to be measured at 3 time points
change in blood brain barrier disruption | baseline, postoperative day 0, postoperative day 1
  biomarker of blood brain barrier disruption to be measured at 3 time points
change in neuronal injury | baseline, postoperative day 0, postoperative day 1
  biomarker of neuronal injury to be measured at 3 time points

SECONDARY OUTCOMES:
delirium as screened with CAM-ICU | twice daily after surgery until discharge from ICU (12 hours, 24 hours, 36 hours, 48 hours, 60 hours, 72 hours, 84 hours, 96 hours, continuing every 12 hours up to 24 weeks)
  CAM-ICU measured twice daily by research assistant to screen for delirium

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States